CLINICAL TRIAL: NCT02149576
Title: Does Intense Regimented Surveillance Improve the Rates of Therapeutic Re-Intervention After Lung Cancer Surgery: A Pilot Study for the Intense-CT Trial
Brief Title: Does Intense Regimented Surveillance Improve the Rates of Therapeutic Re-Intervention After Lung Cancer Surgery
Acronym: Intense-CT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: McMaster Surgical Associates (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: SJHH_IntenseCT_Pilot
Record Dates: First submitted 2014-05-20; First posted 2014-05-29 (Estimated); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Lung Neoplasms
Keywords: Retrospective Review; Pilot Study; Early Stage NSCLC; Post-Surgical Surveillance; Re-intervention Rates
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LDCT Surveillance Program Group (Active Comparator): This cohort will follow a strict schedule of Low Dose Computed Tomography Imaging scans and clinical visits 3, 6, and 12 months after surgery. At each encounter, a history, physical examination, and review of the LDCT results will be performed. Patients with normal clinical and imaging findings will proceed to the next scheduled clinical encounter. Patients with abnormal findings will be managed according to predetermined algorithms.
  Interventions: Procedure: Low Dose Computed Tomography Imaging
- Historical Control Group (Other): The control group will be a retrospective cohort taken from 1-year before the implementation of the LDCT surveillance program. The post-operative follow-up of these participants was not standardized, but rather left up to the discretion of the individual surgeons, and involved chest radiograph imaging as opposed to Low Dose Computed Tomography.
  Interventions: Procedure: Chest Radiograph Imaging

INTERVENTIONS:
Procedure: Low Dose Computed Tomography Imaging
  Arms: LDCT Surveillance Program Group
Procedure: Chest Radiograph Imaging
  Arms: Historical Control Group

SUMMARY:
After curative lung cancer surgery, there is a risk of recurrence of the primary cancer, or development of a new cancer. Historically, patients who have undergone curative lung cancer surgery have been monitored with chest radiographs (CXR). Unfortunately, 70% of such patients still die of lung cancer. As a result, there has been interest in other methods of surveillance in order to detect recurring or new cancers earlier and have more success in treating them. One such technique is Low Dose Computed Tomography (LDCT), which is currently the standard of care and surveillance at this institution. This pilot study aims to determine whether regimented, intensive, short interval LDCT surveillance leads to higher rates of detection and treatment of recurring lung cancers. The study group will be followed up according to a regimented surveillance program using LDCT. The study group will be compared to a group of historical controls whose follow up after surgery was not standardized, but rather left up to the discretion of the individual surgeon. If the results of this study show improvements in detection and treatment of recurrent cancers, it will allow for a larger trial to study the effects of the LDCT surveillance program on lung cancer survival.

The study question aims to determine whether for survivors after curative surgery for Stage I and Stage II lung cancer, a structured Surveillance Program with Low Dose CT can increase the rate of detection and treatment of recurring or new cancers when compared to historical non-structured surveillance with CXR. This study will also determine if it is warranted to pursue a larger scale randomized controlled trial to further investigate optimal LDCT surveillance follow-up intervals and long-term lung cancer survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at minimum 18 years of age
* Patients must have undergone complete resection for pathological Stage I or Stage II lung cancer
* Patients must demonstrate the ability to understand English
* Patients must be able to demonstrate aptitude and willingness to comply with describes study procedures

Exclusion Criteria:

* Patients with residual gross or microscopic disease after surgery
* Patients with pathological Stage III or Stage IV lung cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Rate of therapeutic re-intervention within the first year after curative resection of lung cancer | One year after surgery
  Defined by: 1) rate of curative intent radiation treatment after detection of recurrent or new primary lung cancer 2) rate of curative intent reoperation after detection of recurrent or new primary lung cancer. Measured by frequency of events.

SECONDARY OUTCOMES:
Rate of adherence to follow-up visits | One year after surgery
  Measured by frequency of events
Morbidity of associated interventions | One year after surgery
  Measured by frequency of events

CONTACTS AND LOCATIONS:
Overall Officials: Wael C Hanna, MDCM MBA FRCSC FCCP, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No